CLINICAL TRIAL: NCT06686082
Title: Effectiveness of Biologics on Synovitis and Enthesitis Using Musculoskeletal Ultrasound Assessment in Subclinical Psoriatic Arthritis: a 12-week Observational Real-world Study
Brief Title: A Real-World Study of Biologic Therapy for Subclinical Psoriatic Arthritis
Status: Enrolling by invitation | Type: Observational
Sponsor: Chao Ji (Other)
Responsible Party: Sponsor-Investigator, Chao Ji, professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: FirstAHFujian666
Record Dates: First submitted 2024-11-10; First posted 2024-11-13 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Subclinical Psoriatic Arthritis
Keywords: synovitis; enthesitis
MeSH Terms: conditions — Synovitis | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Subclinical psoriatic arthritis detected by musculoskeletal ultrasound in patients with moderate to severe plaque psoriasis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subclinical psoriatic arthritis patients
  Interventions: Drug: Biologics

INTERVENTIONS:
Drug: Biologics — The ultrasonic changes of synovitis and enthesitis were observed after 12 weeks of treatment with biologic agents

SUMMARY:
Psoriatic arthritis (PsA) is one of the most common comorbidities in patients with psoriasis (PsO). Current research suggests that the progression from PsO to PsA can be divided into five stages of the disease: PsO, preclinical PsA, subclinical PsA, prodromal PsA, and clinical PsA. Subclinical PsA refers to psoriasis participants who do not exhibit any clinical symptoms of arthritis but show evidence of synovio-enthesitis on ultrasound (US). However, there is currently no definitive biomarker that can accurately predict the progression from PsO to PsA. Synovitis and enthesitis are considered important features of PsA. Musculoskeletal ultrasound, using B-mode ultrasound and power Doppler (PD), can visualize synovitis and enthesitis, allowing for the early detection of subclinical PsA, as confirmed by multiple studies. Biologics are currently widely used in the treatment of PsA, with current treatment interventions primarily focusing on patients already diagnosed with PsA. In this study, we conducted a rigorous screening process to identify potential subclinical PsA patients among those with moderate to severe psoriasis. We treated these subclinical PsA patients with biologics and used musculoskeletal ultrasound as a method of efficacy assessment to observe the improvement of synovitis and enthesitis in subclinical PsA patients after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* diagnosed with moderate to severe plaque psoriasis
* no inflammatory arthritis manifestations
* Psoriasis Epidemic Severity Tool (PEST) score ≤ 2
* negative rheumatoid factor
* no prior use of any biologic treatments for psoriasis
* abnormal findings on musculoskeletal ultrasound screening

Exclusion Criteria:

* a previous diagnosis of any other type of arthritis, including rheumatoid arthritis, osteoarthritis, gouty arthritis, ankylosing spondylitis, or similar conditions
* patients with contraindications to the use of biologics
* pregnant or breastfeeding women, and women of childbearing potential who do not agree to use contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate-to-severe plaque psoriasis coming to our hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Improvement of synovitis and enthesitis after 12 weeks of treatment with biological agents. | From enrollment to the end of treatment at 12 weeks
  The assessment using ultrasound was performed at two time points: baseline (0 weeks) and 12 weeks after medication initiation. The joint examination sites were based on the PsAson22. The examination sites for enthesitis were based on the Leeds Enthesitis Index (LEI). According to the European League Against Rheumatism (EULAR)- the Outcome Measures in Rheumatology (OMERACT) definition, the 22 joints with synovitis were scored using ultrasound composite semi-quantitative scale. Additionally, the 6 sites of entheses were evaluated according to the OMERACT enthesitis composite semi-quantitative scale. When assessing joint synovitis and enthesitis using grey scale (GS) and power Doppler (PD), we take the higher score as the final score for that site (range 0 to 3). The total score is the sum of the scores for each site, ranging from 0 to 84.
  Assess the improvement of Sub-PsA patients by evaluating changes before and after treatment through the scoring of synovitis and enthesitis.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No